CLINICAL TRIAL: NCT06659536
Title: Post-market Prospective Clinical Investigation on the Symptomatic Treatment of Urge Incontinence in Adults With Overactive Bladder With Cefar URO
Brief Title: Cefar URO - Symptomatic Treatment of Overactive Bladder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DJO UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENOVIS-S-INP-0003
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-10

CONDITIONS: Overactive Bladder (OAB); Refractory Overactive Bladder; Urinary Urgency and Frequency
Keywords: Urinary urgency; Overactive Bladder (OAB); Transcutaneous Tibial Nerve Stimulation (TTNS); Cefar Uro
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous Tibial Nerve Stimulator (TTNS) with the Cefar Uro Device (Experimental): Patients will undergo Transcutaneous Posterior Tibial Nerve Stimulation with the Cefar URO device. The following parameters setting (preset program P4) will be used for treatment of all enrolled subjects:
  * frequency of 20Hz
  * pulse width of 200 μs
  * duration: 30 minutes per treatment.
  * treatment frequency: subjects will be recommended to have 7 treatment sessions per week for a total of 12 weeks (84 treatments total), and anyway no less that one treatment per week.
  The electrodes will be placed in the medial ankle as according to the device IFU.
  Interventions: Device: Transcutaneous Tibial Nerve Stimulation (TTNS) with the Cefar Uro Device

INTERVENTIONS:
Device: Transcutaneous Tibial Nerve Stimulation (TTNS) with the Cefar Uro Device — Transcutaneous Tibial Nerve Stimulation (TTNS) with the Cefar URO device using the preset program P4 (parameter setting: frequency 20Hz, pulse width 200μs) for the symptomatic treatment of urge incontinence in adults with overactive bladder in accordance with the approved labelling.

SUMMARY:
A Post-Market Prospective Clinical Investigation to collect PMCF data on the safety and performance of the Cefar URO device when using the preset program P4 (parameter setting: frequency 20Hz, pulse width 200μs) for the symptomatic treatment of urge incontinence in adults with overactive bladder in accordance with the approved labelling.

The Cefar URO device features four pre-set programs (P1, P2, P3 and P4) and three custom programs. Although supporting data on the preset programs P1, P2, P3 are available for the clinically equivalent UROstim2 device, program P4 is unique to Cefar URO. Program P4 utilizes the parameters 20Hz and 200μs which are commonly reported in the literature for the stated indications but for which no data is available for the clinically equivalent UROstim2 device. The present study is therefore aimed to cover this data gap.

DETAILED DESCRIPTION:
The objectives of this prospective study are to assess the performance and safety of Cefar URO when used at home by enrolled patients using the P4 program pre-set parameters i.e. frequency 20Hz, pulse width 200μs, for 12 weeks.

Adult patients who require symptomatic treatment of urge incontinence and associated symptoms with overactive bladder (including refractory overactive bladder of idiopathic or neurogenic origin), will undergo Transcutaneous Posterior Tibial Nerve Stimulation with the Cefar URO device at home.

The diagnosis of OAB is made by the Investigator on the basis of clinical symptoms in routine practice.

The assessment of symptoms and quality of life of patients will be completed before treatment (Baseline) and after 6 and 12 weeks of treatment with the Cefar URO device. An additional assessment of the maintenance of symptoms and quality of life will be performed 4 weeks after end of the per protocol treatment.

The tests used to assess symptoms and quality of life are and compliance with treatment are:

1. the Overactive bladder Questionnaire (OAB-q) SF 4 Weeks Recall (6-item Symptom Bother Scale and a 13-item HRQL Scale)
2. the 3-day bladder diary
3. A 6-point Likert scale to assess faecal incontinence (only in case patients experience faecal incontinence at baseline)
4. Compliance diary

The following parameters setting (preset program P4) will be used for treatment of all enrolled subjects with the Cefar URO device:

* frequency of 20Hz
* pulse width of 200 μs
* duration: 30 minutes per treatment.
* treatment frequency: subjects will be recommended to have 7 treatment sessions per week for a total of 12 weeks (84 treatments total), and anyway no less that one treatment per week.

The electrodes will be placed in the medial ankle as according to the device IFU.

Patients will be asked to record each treatment session performed on the patient's diary, in order to assess compliance with the scheduled treatment plan.

The subjects will be treated for a period of 12 weeks with the Cefar URO device as per the treatment protocol described above.

After completion of the per protocol treatment period, the subjects will be followed up for an additional period of 4 weeks. During these four weeks, patients will be asked to continue performing the treatment according to their needs and according to the Investigator's instructions (Maintenance treatment protocol). No prescription about the number of treatments is imposed by the protocol during this period.

The subjects will be evaluated at study site for 6 on site visits and 10 weekly phone contacts, as detailed in the study flowchart at the end of this section.

Weekly follow-up phone contacts with the patients will be performed during the 12 weeks of the per protocol treatment with the exception of the weeks when an onsite visit is scheduled. One additional phone call will be performed during the exploratory long term 4 weeks follow up period (Maintenance period). These regular contacts serve to remind the patient to follow the treatment plan and to complete the self-reported questionnaires accurately. Additionally, at each phone contact patients will be asked to report if any issues/adverse events have been occurred since the last visit or phone contact. The regular phone contact with patients should help in keeping the adherence to the protocol and have a higher compliance to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with overactive bladder (including refractory overactive bladder of idiopathic or neurogenic origin) who require symptomatic treatment of urge incontinence and associated symptoms.
* Subjects, both male and female, ≥ 18 years of age at the time of consent
* Subjects have provided their written consent to participate in the study by signing the Ethics-approved consent form.
* Patients are considered able and willing to self-administer transcutaneous tibial nerve stimulator (TTNS) treatment at home, based on Investigator's judgement.
* Patients are suitable to receive treatment using the Cefar URO device P4 program pre-set parameters (frequency 20Hz and pulse width 200μs) for 12 weeks, based on Investigator's judgement.
* If undergoing pharmacological therapy for incontinence, the therapy must be stabilized for at least 4 weeks before baseline visit

Exclusion Criteria:

* Pregnancy confirmed by urine test at screening
* Urinary tract infection confirmed by urine analysis
* Serious secondary illness (such as renal failure, nephrolithiasis, bladder and kidney tumors)
* Detrusor-sphincter dyssynergia
* Patients who have or have had implantable neurostimulating cardiac demand pacemakers, ICD; or other implantable electronic devices
* Subjects who are not able to read and understand the Instructions for Use, warnings, cautions and dangers
* Subjects who are not able to read and understand indications and contraindications of the device
* Subjects who are not able to sense auditory and visual signals
* Patients with anti-incontinence surgery planned during the course of the study
* Participation in another clinical study within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From enrollment to the end of Treatment at 16 weeks.
  - adverse events/malfunctions/complications reported during the study. Subjects and Investigators will be prompted to record such issues on the AE evaluation form.
Frequency of Overactive Bladder Symptoms | From enrollment to the end of Treatment at 12 weeks.
  - change in symptoms, at 12 weeks, quantified as the mean change from baseline on the Overactive Bladder-questionnaire-Short Form (OAB-q-SF), Symptoms bother scale (6 items) based on patient self-reporting.
  The lowest score for symptoms is 6, and the highest is 36. Higher score values are indicative of grater symptom bother and lower scores indicate minimal symptom bother.
  As per the literature (Zonic-Imamovic et al.,2021), we may expect an approximate mean reduction of the Symptoms Bother scale of 10.4 points at 12 weeks compared to the baseline measurement.

SECONDARY OUTCOMES:
Number of Urinary Urgency and Urinary Frequency Episodes | From enrollment to the end of Treatment at 12 weeks.
  - change in the number of episodes of Urinary Urgency and Urinary Frequency measured at 12 weeks compared to baseline, measured by means of 3-day bladder patient diary. This will quantify the average number of urgency and frequency episodes per day over three consecutive days, allowing for a direct comparison of baseline and 12-week data.
Change in Quality of Life | From enrollment to the end of Treatment at 12 weeks.
  - change in Health-Related Quality of Life as shown by a reduction in the Overactive Bladder-questionnaire-Short Form (OAB-q-SF), Health-Related Quality of Life (HRQoL) (13 items) at 12 weeks relative to baseline, based on patient self reported outcomes.
  To assess the quality of life, the lowest score is 13 and the highest is 78. Higher scores will be indicative of better HRQL.

OTHER OUTCOMES:
Number of Urinary Incontinence and Nocturia episodes | From enrollment to the end of Treatment at 12 weeks.
  - change in the number of episodes of Urinary Incontinence and Nocturia, assessed at 12 weeks compared to baseline using a 3-day bladder diary. This endpoint will quantify the average daily episodes for both incontinence and nocturia across three consecutive days, enabling a direct comparison of baseline and 12-week data.
Frequency of Overactive Bladder Symptoms at a longer term follow up | From enrollment to the end of Treatment at 16 weeks.
  - Maintenance of Symptoms Bother between 12 and 16 weeks, assessed using the Symptoms Bother Scale from the Overactive Bladder-questionnaire-Short Form (OAB-q-SF). Maintenance will be defined as no statistically significant worsening in symptom-related distress between 12 and 16 weeks.
  The lowest score for symptoms is 6, and the highest is 36. Higher score values are indicative of grater symptom bother and lower scores indicate minimal symptom bother.
Change in Quality of Life at a longer term follow up | From enrollment to the end of Treatment at 16 weeks.
  - maintenance of Health-Related Quality of Life (HRQoL) between 12 and 16 weeks, measured using the HRQoL component of the Overactive Bladder-questionnaire-Short Form (OAB-q-SF). Maintenance will be defined as no statistically significant worsening in HRQoL scores over this period.
  To assess the quality of life, the lowest score is 13 and the highest is 78. Higher scores will be indicative of better HRQL.
Frequency of Overactive Bladder Symptoms and Change in Quality of Life at a longer term follow up | From enrollment to the end of Treatment at 16 weeks.
  - Maintenance of urinary symptom severity between 12 and 16 weeks, measured using the 3-day bladder diary. Maintenance will be defined as no statistically significant increase in the average daily episodes of Urinary Urgency, Frequency, Incontinence, and Nocturia over three consecutive days..
Change in symptoms of faecal incontinence | From enrollment to the end of Treatment at 12 weeks.
  Change in faecal incontinence symptoms during the treatment period, assessed for patients who report faecal incontinence at baseline. Symptom change will be measured using a 6-point Likert scale (where 1 means "condition resolved" and 6 "condition significanty worsen") at 12 weeks, with analysis exploring whether peripheral neuromodulation yields a positive effect on urge faecal incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, Pr., Principal Investigator — Service de Neuro-Urologie, Hôpital Tenon
Locations (1):
- Neuro-Urology Department, Tenon Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No